CLINICAL TRIAL: NCT00271843
Title: Predicting Tobacco and Alcohol Initiation
Brief Title: Smoking and Alcohol Initiation
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Other Study IDs: 1R21DA019916-01 (NIH)
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2008-12

CONDITIONS: Smoking; Alcohol Drinking
MeSH Terms: conditions — Smoking; Alcohol Drinking

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study evaluates multi-attribute utility, a modification of subjective expected utility, as a descriptive model of the adolescent's decision to initiate smoking or alcohol use. According to the model, the young decision maker envisions a set of consequences that will follow the two decision options, either to continue as a non-user or to initiate usage. Each consequence has three components. The components are the worth of the consequence, which may be positive or negative, the judged likelihood that the consequence will happen, and the importance of the consequence. Within an individual, importances will change with mood or circumstance, which is how the model accounts for impulsive decisions that may occur in social settings.

The model will be tested by eliciting components of ten independent consequences from a large group of students early in the seventh-grade year. Current usage will also be examined; extant data suggest that most students will be non-users at that time. It is known that a fair amount of initiation takes place during the seventh and eighth grade years. The hypothesis is that those non-users whose model scores are high will be more likely to initiate usage than those whose scores are low. The same students will be queried regarding usage eighteen months later to evaluate the hypothesis.

It is now well known that differential knowledge regarding the harmful effects of drug use does not distinguish adolescent users from non-users. The model approach quantifies the idea that anticipated positive consequences play a prominent role in the decision of those who choose to initiate. An important implication is that prevention campaigns might profit by addressing positive as well as negative consequences of usage.

DETAILED DESCRIPTION:
A book entitled "A science of decision making: the legacy of Ward Edwards" and 4 chapters were published (Oxford University Press, 2008) with the support of this funding.

ELIGIBILITY:
Inclusion Criteria:

* enrolled middle school students

Exclusion Criteria:

* N/A

Ages: 11 Years to 15 Years | Sex: All
Age Groups: Child
Enrollment: 2600 (Estimated)
Dates: Start 2005-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jie W. Weiss, Ph.D., Principal Investigator — California State University, Fullerton
Locations (1):
- California State University, Fullerton, California, United States

REFERENCES:
- [Background] Weiss, J. W., & Weiss, D. J. (Eds.) (in press). The essential Ward Edwards. New York: Oxford University Press.
- [Background] Weiss, J. W., & Edwards, W., Mouttapa, M. (in press). The puzzle of adolescent substance initiation. In J. W. Weiss & D. J. Weiss (Eds). The essential Ward Edwards. New York: Oxford University Press.
- [Background] Weiss, J. W., Weiss, D. J., & Edwards, W. (in press). Big decisions, little decisions: The hierarchy of everyday life. In J. W. Weiss & D. J. Weiss (Eds). The essential Ward Edwards. New York: Oxford University Press.